CLINICAL TRIAL: NCT03197766
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of BMN 111 in Children With Achondroplasia
Brief Title: A Study to Evaluate the Efficacy and Safety of BMN 111 in Children With Achondroplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111-301; 2015-003836-11 (EudraCT Number)
Record Dates: First submitted 2017-05-23; First posted 2017-06-23 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Achondroplasia
Keywords: Achondroplasia; Dwarfism; Bone Diseases; Bone Diseases, Developmental; ACH; Natriuretic Peptide, C-Type; Musculoskeletal Diseases; Natriuretic Agents; Physiological Effects of Drugs; Skeletal Dysplasias; Genetic Diseases, Inborn; Osteochondrodysplasias
MeSH Terms: conditions — Achondroplasia; Dwarfism; Bone Diseases; Bone Diseases, Developmental; Musculoskeletal Diseases; Genetic Diseases, Inborn; Osteochondrodysplasias | interventions — vosoritide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Active BMN 111 (Experimental): Daily subcutaneous injection of 15 micrograms per kilogram BMN111
  Interventions: Drug: BMN 111
- Placebo (Placebo Comparator): Daily subcutaneous injection of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMN 111 — Subcutaneous injection of 15 μg/kg of BMN 111 daily
  Other Names: Vosoritide; Modified recombinant human C-type natriuretic peptide
  Arms: Active BMN 111
Drug: Placebo — Subcutaneous injection of 15 μg/kg of placebo daily
  Arms: Placebo

SUMMARY:
The intent and design of this Phase 3 study is to assess BMN 111 as a therapeutic option for the treatment of children with Achondroplasia.

DETAILED DESCRIPTION:
This is a Phase 3 randomized, placebo-controlled, double-blind multicenter study with approximately 110 subjects, aged 5 to < 18 years old. Subjects with documented Achondroplasia confirmed by genetic testing will have been enrolled in Study 111-901 for at least a 6-month period immediately before entering into the 111-301 study. Eligible subjects will be randomly assigned to one of two treatment groups: placebo or BMN 111 at 15 μg/kg. The route of administration is subcutaneous injection and the frequency is daily.

ELIGIBILITY:
Inclusion Criteria

* Parent(s) or guardian(s) consent
* 5 to < 18 years old
* ACH, documented and confirmed by genetic testing
* At least a 6-month period of pretreatment growth assessment in Study 111-901 before study entry
* If sexually active, willing to use a highly effective method of contraception
* Ambulatory and able to stand without assistance

Exclusion criteria:

* Hypochondroplasia or short stature condition other than ACH
* Have any of the following:

  * Hypothyroidism or hyperthyroidism
  * Insulin-requiring diabetes mellitus
  * Autoimmune inflammatory disease
  * Inflammatory bowel disease
  * Autonomic neuropathy
* History of any of the following:

  * Renal insufficiency defined as serum creatinine > 2 mg/dL
  * Chronic anemia
  * Baseline systolic blood pressure (BP) < 70 millimeters of mercury (mm Hg) or recurrent symptomatic hypotension (defined as episodes of low BP generally accompanied by symptoms ie, dizziness, fainting) or recurrent symptomatic orthostatic hypotension
  * Cardiac or vascular disease

    * Have a clinically significant finding or arrhythmia on screening electrocardiogram (ECG) that indicates abnormal cardiac function or conduction or Fridericias corrected QTc-F > 450 msec
* Have an unstable condition likely to require surgical intervention during the study (including progressive cervical medullary compression or severe untreated sleep apnea)
* Decreased growth velocity (< 1.5 cm/yr) over a period of 6 months or evidence of growth plate closure (proximal tibia, distal femur)
* Treated with growth hormone, insulin-like growth factor 1 (IGF-1), or anabolic steroids in the previous 6 months or treatment greater than 6 months at any time
* Greater than 1 month treatment with oral corticosteroids (low-dose ongoing inhaled steroid for asthma, or intranasal steroids, are acceptable) in the previous 12 months
* Planned or expected to have limb-lengthening surgery during the study period. Subjects with previous limb- lengthening surgery may enroll if surgery occurred at least 18 months prior to the study and healing is complete without sequelae.
* Planned or expected bone-related surgery (ie. surgery involving disruption of bone cortex, excluding tooth extraction), during the study period. Subjects with previous bone-related surgery may enroll if surgery occurred at least 6 months prior to the study and healing is complete without sequelae.
* Had a fracture of the long bones or spine within 6 months prior to screening
* History of severe untreated sleep apnea
* New initiation of sleep apnea treatment (e.g. CPAP or sleep apnea-mitigating surgery) in the previous 2 months prior to screening
* History of hip surgery or hip dysplasia atypical for achondroplastic subjects
* History of clinically significant hip injury in the 30 days prior to screening
* History of slipped capital femoral epiphysis or avascular necrosis of the femoral head
* Abnormal findings on baseline clinical hip exam or imaging assessments that are determined to be clinically significant
* Concurrent disease or condition that would interfere with study participation or safety evaluations, for any reason
* Condition or circumstance that places the subject at high risk for poor treatment compliance or for not completing the study

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 121 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (24):
- United States (11):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Emory University, Decatur, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of Missouri, Columbia, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Children's Hospital, Milwaukee, Wisconsin
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Murdoch Children's Research Institute, Parkville, Victoria
- Germany (2):
  - Otto-von-Guericke Universitaet, Universitaetskinderklinik, Magdeburg
  - Universitätsklinikum Münster, Münster
- Japan (3):
  - Osaka University Hospital, Osaka
  - Saitama Children's Medical Center, Saitama
  - Tokushima University Hospital, Tokushima
- Spain (3):
  - Institut Catala de Traumatologica I Medicina de l'Esport, Barcelona
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario Virgen de la Victoria, Málaga
- Acibadem University School of Medicine, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Guy's and St. Thomas NHS Foundation Trust Evelina Children's Hospital, London
  - Sheffield Children's NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Savarirayan R, Irving M, Wilcox WR, Bacino CA, Hoover-Fong JE, Harmatz P, Polgreen LE, Palm K, Prada CE, Kubota T, Arundel P, Kotani Y, Leiva-Gea A, Bober MB, Hecht JT, Legare JM, Lawrinson S, Low A, Sabir I, Huntsman-Labed A, Day JRS. Sustained growth-promoting effects of vosoritide in children with achondroplasia from an ongoing phase 3 extension study. Med. 2025 May 9;6(5):100566. doi: 10.1016/j.medj.2024.11.019. Epub 2024 Dec 30. PMID 39740666
- [Derived] Savarirayan R, Irving M, Wilcox WR, Bacino CA, Hoover-Fong JE, Harmatz P, Polgreen LE, Mohnike K, Prada CE, Kubota T, Arundel P, Leiva-Gea A, Rowell R, Low A, Sabir I, Huntsman-Labed A, Day J. Persistent growth-promoting effects of vosoritide in children with achondroplasia are accompanied by improvements in physical and social aspects of health-related quality of life. Genet Med. 2024 Dec;26(12):101274. doi: 10.1016/j.gim.2024.101274. Epub 2024 Sep 18. PMID 39305160
- [Derived] Qi Y, Chan ML, Mould DR, Larimore K, Fisheleva E, Cherukuri A, Day J, Savarirayan R, Irving M, Bacino CA, Hoover-Fong J, Ozono K, Mohnike K, Wilcox WR, Bober MB, Henshaw J. Development of a Weight-Band Dosing Approach for Vosoritide in Children with Achondroplasia Using a Population Pharmacokinetic Model. Clin Pharmacokinet. 2024 May;63(5):707-719. doi: 10.1007/s40262-024-01371-6. Epub 2024 Apr 23. PMID 38649657
- [Derived] Chan ML, Qi Y, Larimore K, Cherukuri A, Seid L, Jayaram K, Jeha G, Fisheleva E, Day J, Huntsman-Labed A, Savarirayan R, Irving M, Bacino CA, Hoover-Fong J, Ozono K, Mohnike K, Wilcox WR, Horton WA, Henshaw J. Pharmacokinetics and Exposure-Response of Vosoritide in Children with Achondroplasia. Clin Pharmacokinet. 2022 Feb;61(2):263-280. doi: 10.1007/s40262-021-01059-1. Epub 2021 Aug 25. PMID 34431071
- See also: NIH Genetics Home Reference related topics: Achondroplasia — https://ghr.nlm.nih.gov/condition/achondroplasia
- See also: NIH Genetic and Rare Diseases Information Center resources: Achondroplasia — https://rarediseases.info.nih.gov/diseases/8173/achondroplasia
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-centre study conducted by 24 principal investigators at 24 study centers in 7 countries
Pre-assignment Details: A total of 121 subjects were enrolled into the study, 119 subjects completed and 2 subjects withdrew from the study.
Groups:
- BMN 111 - 15 μg/kg: BMN 111: Subcutaneous injection of 15 μg/kg of BMN 111 daily
- Placebo: Placebo: Subcutaneous injection of placebo daily
Period: Overall Study
Arm/Group | BMN 111 - 15 μg/kg | Placebo
Started | 60 | 61
Completed | 58 | 61
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Analysis were performed on the Full Analysis Set (FAS) which included all randomized subjects with a signed informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | BMN 111 - 15 μg/kg | Placebo | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.35 (2.43) | 9.06 (2.47) | 8.71 (2.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 31 | 33 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 7
  Not Hispanic or Latino | 59 | 55 | 114
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 45 | 41 | 86
  Race: Asian-Other | 7 | 9 | 16
  Race: Asian-Japanese | 3 | 4 | 7
  Race: Multiple | 2 | 5 | 7
  Race: Black or African American | 3 | 2 | 5
Annualized Growth Velocity (AGV) [Mean (Standard Deviation); unit: cm/year] | 4.26 (1.53) | 4.06 (1.20) | 4.16 (1.37)
Height Z-Score [Mean (Standard Deviation); unit: Z-score] — A height Z score of 0 would indicate that the subject's height is equal to the mean height for the average stature population of the same sex and age.
  Z-score | -5.13 (1.11) | -5.14 (1.07) | -5.13 (1.09)
Upper to Lower Body Segment Ratio [Mean (Standard Deviation); unit: Ratio] | 1.98 (0.20) | 2.01 (0.21) | 2.00 (0.20)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Annualized Growth Velocity (AGV) at Week 52
Description: AGV at a Post-baseline Visit is defined as [(Height at Post-baseline Visit - Height at Baseline)/(Date of Post-baseline Visit - Date of Baseline Assessment)] x 365.25
  AGV at Baseline is defined as [(Height at Baseline - last height measurement in Study 111-901 at least 6 months prior to Baseline)/(Date of Baseline Assessment - Date of last height measurement in Study 111-901 at least 6 months prior to Baseline)] x 365.25
Time Frame: At Baseline and Week 52
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: cm/year
Arm/Group | BMN 111 - 15 μg/kg | Placebo
Number analyzed (Participants) | 60 | 61
cm/year | 1.71 [1.40 to 2.01] | 0.13 [-0.18 to 0.45]
Statistical Analysis 1: Comparison: BMN 111 - 15 μg/kg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Confirmatory statistical testing controlling for the Type I error rate was performed on the primary analysis for the primary endpoint; Two subjects in the BMN 111 group discontinued from the study before Week 52. The values for these 2 subjects were imputed for this analysis

2. Secondary Outcome: Change From Baseline in Height Z-score at Week 52
Description: Z-Scores were derived using age-sex specific reference data (means and SDS) for average stature children per the Centers for Disease Control and Prevention.
  A height Z score of 0 would indicate that the subject's height is equal to the mean height for the average stature population of the same sex and age.
  A positive height Z score indicates that the subjects height is above the mean height for the average stature population of the same sex and age, whilst a negative height Z score indicates that the subjects height is below the mean height for the average stature population of the same sex and age.
  To conclude if the height Z score increases then this means the height deficit has decreased.
Time Frame: At baseline and Week 52
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Z-Score
Arm/Group | BMN 111 - 15 μg/kg | Placebo
Number analyzed (Participants) | 60 | 61
Z-Score | 0.27 [0.18 to 0.36] | -0.01 [-0.10 to 0.09]
Statistical Analysis 1: Comparison: BMN 111 - 15 μg/kg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Confirmatory statistical testing controlling for the Type I error rate was performed on the primary analyses for the two key secondary endpoints; Missing assessments at Week 52 were imputed

3. Secondary Outcome: Change From Baseline in Upper to Lower Segment Body Ratio at Week 52
Description: Evaluate change from baseline in mean upper:lower segment body ratio in subjects treated with BMN 111 compared with control subjects in the placebo group at 52 weeks
Time Frame: At baseline and Week 52
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | BMN 111 - 15 μg/kg | Placebo
Number analyzed (Participants) | 60 | 61
Ratio | -0.03 [-0.06 to 0.00] | -0.02 [-0.05 to 0.01]
Statistical Analysis 1: Comparison: BMN 111 - 15 μg/kg vs Placebo; Test type: Superiority; p = 0.506, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Missing assessments at Week 52 were imputed

4. Secondary Outcome: Summary of Subjects Experiencing Adverse Events (AEs) During Treatment
Description: AEs with onset or worsening after the initiation of study drug and up to 30 days after study drug discontinuation were included.
  serious adverse event (SAE)
Time Frame: Up to Week 56
Population: The Safety Population was defined as all subjects in the FAS who received at least one dose of double-blind BMN 111 or placebo in this study.
Measure: Number; unit: participants
Arm/Group | BMN 111 - 15 μg/kg | Placebo
Number analyzed (Participants) | 60 | 61
participants
  Subjects with any AE | 59 | 60
  Subjects with any SAE | 3 | 4
  Subjects with any treatment-related AE | 53 | 51
  Subjects who died | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 56
Description: A treatment-emergent Adverse Event (TEAE) is any Adverse Event with onset or worsening after the initiation of study drug and up to 30 days after study drug discontinuation were included. The Safety Population is defined as all subjects in the FAS who received at least one dose of double-blind BMN 111 or placebo in this study
Arm/Group | BMN 111 - 15 μg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/61
Serious Adverse Events (participants affected / at risk) | 3/60 | 4/61
Other Adverse Events (participants affected / at risk) | 59/60 | 60/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMN 111 - 15 μg/kg (N=60) | Placebo (N=61)
Influenza (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMN 111 - 15 μg/kg (N=60) | Placebo (N=61)
Injection site reaction (General disorders) | 44 | 29
Injection site erythema (General disorders) | 41 | 40
Injection site swelling (General disorders) | 23 | 6
Pyrexia (General disorders) | 10 | 13
Injection site urticaria (General disorders) | 8 | 2
Injection site bruising (General disorders) | 5 | 8
Fatigue (General disorders) | 4 | 0
Injection site mass (General disorders) | 4 | 1
Injection site rash (General disorders) | 3 | 0
Injection site haemorrhage (General disorders) | 2 | 7
Injection site induration (General disorders) | 2 | 0
Injection site inflammation (General disorders) | 2 | 1
Injection site pain (General disorders) | 2 | 5
Injection site vesicles (General disorders) | 2 | 3
Gait disturbance (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Injection site discolouration (General disorders) | 1 | 2
Injection site pruritus (General disorders) | 1 | 4
Malaise (General disorders) | 1 | 2
Pain (General disorders) | 1 | 0
Feeling hot (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 0 | 1
Medical device pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Secretion discharge (General disorders) | 0 | 1
Vaccination site reaction (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 16 | 18
Upper respiratory tract infection (Infections and infestations) | 8 | 10
Ear infection (Infections and infestations) | 6 | 6
Influenza (Infections and infestations) | 5 | 3
Otitis media (Infections and infestations) | 6 | 6
Viral infection (Infections and infestations) | 5 | 3
Gastroenteritis (Infections and infestations) | 4 | 3
Gastroenteritis viral (Infections and infestations) | 4 | 1
Tonsillitis (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 2 | 1
Enterobiasis (Infections and infestations) | 2 | 0
Otitis externa (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 1
Impetigo (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Otitis media acute (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 4
Scarlet fever (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 2
Streptococcal infection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 2
Fungal skin infection (Infections and infestations) | 0 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 1
Lice infestation (Infections and infestations) | 0 | 2
Molluscum contagiosum (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 14 | 16
Dizziness (Nervous system disorders) | 4 | 1
Paraesthesia (Nervous system disorders) | 2 | 1
Presyncope (Nervous system disorders) | 2 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Hyperreflexia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Extensor plantar response (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 2
Poor quality sleep (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 16 | 12
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Gingival pain (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Malpositioned teeth (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Anal pruritus (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 2
Oral pain (Gastrointestinal disorders) | 0 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 3 | 2
Bone contusion (Injury, poisoning and procedural complications) | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1
Procedural anxiety (Injury, poisoning and procedural complications) | 2 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 6 | 3
Otorrhoea (Ear and labyrinth disorders) | 3 | 3
Tympanic membrane perforation (Ear and labyrinth disorders) | 2 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 1
Excessive cerumen production (Ear and labyrinth disorders) | 1 | 0
External ear inflammation (Ear and labyrinth disorders) | 1 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Blood pressure decreased (Investigations) | 7 | 3
Body temperature increased (Investigations) | 2 | 0
Seasonal allergy (Immune system disorders) | 4 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Device expulsion (Product Issues) | 1 | 0
Enuresis (Psychiatric disorders) | 1 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Trichotillomania (Psychiatric disorders) | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 1
Defect conduction intraventricular (Cardiac disorders) | 0 | 1
Diastematomyelia (Congenital, familial and genetic disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03197766/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT03197766/SAP_001.pdf